CLINICAL TRIAL: NCT00463580
Title: An Evaluation of the Efficacy of the Tumor Necrosis Factor-alpha Antagonist Infliximab in Treatment Resistant Major Depression: Mechanisms and Mediators
Brief Title: A Study of Infliximab for Treatment Resistant Major Depression
Acronym: Infliximab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00011734; 1R21MH077172-01A2 (NIH)
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: depression; TNF-alpha antagonist; infliximab; treatment resistant depression; major depressive disorder (MDD); bipolar I disorder; bipolar II disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder | interventions — Infliximab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Participants in this arm will receive an infusion of infliximab.
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Participants in this arm will receive an infusion of normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — Participants will receive three infusions 5mg/kg of infliximab (at Baseline, Week 2 and Week 6)
  Other Names: Remicade
  Arms: Infliximab
Drug: Placebo — Participants will receive three infusions of a placebo (at Baseline, Week 2 and Week 6)
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
Major depression is increasingly recognized to be a chronic and highly recurrent condition, which results in significantly increased health problems. One possible mechanism that may contribute to treatment resistance is increased production and release of chemicals called proinflammatory cytokines in patients with major depression. These chemicals mediate the body's response to infectious agents like bacteria and have been shown to be increased by psychological stress. They produce the symptoms that we associate with being sick, including fever, malaise and changes in sleep and appetite. Several lines of evidence indicate that proinflammatory cytokines may contribute to the development of major depression and may thus represent a novel target for the pharmacological treatment of the disorder.

The TNF-alpha antagonist, Infliximab (Remicade®), is an infusion style drug approved by the FDA for the treatment of inflammatory conditions like Crohns disease and rheumatoid arthritis. The researchers are conducting a study to see if the infliximab (Remicade®) is more effective than placebo in acutely reducing symptoms of depression in patients who have elevated proinflammatory markers and have not responded to, or been unable to tolerate, at least two previous treatments in the current depressive episode. Proinflammatory markers are measured by a simple blood test for C-Reactive Protein (CRP) levels in the body.

DETAILED DESCRIPTION:
Major depression has become a health crisis of epidemic proportions in the modern world. The prevalence of major depression has risen over the last several generations in every country examined, and age of symptom onset has decreased. Currently the fourth leading health burden worldwide, major depression will rank second after cardiac disease as a cause of international medical morbidity by the year 2020. One in six individuals in the United States will experience an episode of major depression in his or her lifetime, and the risk of subsequent episodes rises dramatically once a person has been depressed. Indeed, depression is now recognized to be a highly chronic and recurrent illness. On average, patients with major depression are symptomatic 60% of the time, even when receiving community-standard antidepressant treatment. Recent estimates place the economic burden of depression in the United States at 83 billion dollars a year.

Depression is associated with greater disability than are most other chronic illnesses and is a risk factor for mortality. Suicide ranks among the top ten causes of death in the United States, and best estimates suggest that 60-70% of people who kill themselves are clinically depressed. Between 10-15% of severely depressed people eventually commit suicide. In addition, many studies indicate that depression significantly increases all-cause mortality independently of suicide. Depression predicts the later development of a number of medical conditions, including cardiac and cerebrovascular disease, hypertension,diabetes,obesity and the metabolic syndrome,dementia, and cancer. Depression also markedly increases mortality in patients who are medically ill and has been associated with decreased responses to pharmacological treatments for cancer and hepatitis C.

Unfortunately, most patients with depression do not experience a complete resolution of symptoms with antidepressant treatment and 10-20% of patients are refractory to all currently available modalities, including electroconvulsive shock (ECT) therapy. ECT is often effective in patients who have failed adequate trials of multiple antidepressants, but is associated with the risk of anesthesia and with significant short term memory impairment. Responses to ECT are short-lived, and many patients who respond subsequently relapse, even when on maintenance antidepressants. In addition to efficacy issues, many patients are unable to tolerate side effects associated with antidepressants or ECT. The risks of not responding to (or tolerating) treatment have been highlighted by recent studies documenting that partial-but incomplete-response is associated with an increased risk of full symptomatic relapse (even when on therapy) and a worse long term disease course, as well as with significantly impaired quality of life. Treatment resistance also results in a six times increase in direct health care costs. These factors highlight the tremendous need to identify novel treatment strategies, especially for depressed patients who are unresponsive to conventional therapies.

One possible mechanism that may contribute to treatment resistance is increased proinflammatory cytokine production and release. Several lines of evidence indicate that proinflammatory cytokines participate in the pathophysiology of major depression and may thus represent a novel target for the pharmacological treatment of the disorder. First, a high percentage of patients who receive cytokine therapies (such as interferon-alpha for malignant melanoma or hepatitis C infection) develop depressive symptoms, and many patients meet full criteria for major depression. Interferon-alpha-induced depressive symptoms can be ameliorated by pre-treatment with an antidepressant and respond to antidepressants once they have emerged. Second, many studies report that, as a group, medically healthy patients with depression exhibit elevated measures of proinflammatory cytokines, including tumor necrosis factor (TNF)-alpha, interleukin (IL)-1 and IL-6. Moreover, a positive relationship between serum concentrations of proinflammatory cytokines and severity of depressive symptoms has been recently reported. Third, antidepressants have been shown to have anti-inflammatory activity and may work-at least in part-by reducing inflammatory activity, given evidence that clinical response is associated with reductions in cytokine levels. These data raise the possibility that cytokine antagonists, such as the chimeric anti-TNF-alpha antibody infliximab, might have antidepressant efficacy. Of special relevance to this proposal, patients who are treatment resistant have been shown to exhibit increased inflammatory activity (as reflected by increased plasma concentrations of interleukin [IL]-6 and the soluble IL-6 receptor [sIL-6R]), suggesting that cytokine antagonists might be especially effective in these patients.

Providing care to patients with inflammatory bowel disease has given us the clear clinical impression that infliximab rapidly improves mood and energy levels in many patients prior to any demonstrable changes in bowel pathology. This impression is in line with a growing body of evidence suggesting that TNF-alpha antagonists improve emotional functioning and fatigue in patients receiving these agents for rheumatoid arthritis and inflammatory bowel disease. These findings in patients with inflammatory diseases are consistent with the notion that TNF-alpha antagonists such as infliximab might provide acute symptomatic relief for medically healthy patients with treatment-resistant major depression and that symptom improvement might result from decreased inflammatory activity. Moreover, medically healthy depressed patients with increased inflammatory activity may be most likely to benefit from anti-TNF-alpha therapy.

After appropriate screening to determine eligibility, 64 subjects with treatment resistant depression will be randomized to receive three infusions of either infliximab (Remicade®) or placebo (salt water) in the Emory Infliximab Infusion Center in the Division of Digestive Diseases, Emory University School of Medicine. Subjects will be followed for 12 weeks with evaluations at weeks 0 (baseline), 1, 2, 3, 4, 6, 8, 10 and 12. The first infliximab (Remicade®) infusion will occur at the first (Baseline) visit. The second infusion will occur at Study Week 2 (the third visit). The third infusion will occur at Study Week 6 (Visit 6). The choice of three infusions, and the infusion schedule, is based on current recommendations for the use of infliximab (Remicade®) in conditions for which it has received FDA approval. Subjects will be evaluated for twelve weeks by trained clinicians for changes in depression symptoms and improvements in quality of life. In addition, a physician will evaluate subjects each visit to make sure they are remaining healthy. Blood will be drawn at baseline prior to infusion and all subsequent visits to check labs for safety but also to evaluate potential relationships between changes in inflammatory activity and therapeutic response. After Study Week 12, participants will be monitored by phone, every 4 weeks during the 22-Week Post Study Follow-up Phase to assess physical and psychiatric symptoms in the period following the final infusion. At the baseline and Week 8 visits, subjects will be admitted to the Atlanta Clinical Translational Science Institute (ACTSI), a research unit in the Emory Hospital, for an extended evaluation. The purpose of coming to the ACTSI will be for researchers to evaluate whether treatment with infliximab improves endocrine function, inflammation, sleep and thinking abilities in people who are depressed. For all other visits (Week 1, 2, 4, 6, 10 and 12), participants will come for an office visit in the Winship Cancer Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages 25-60. Must be able to read and understand English.
2. Currently meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-IV) criteria for a major depressive episode. (History of either unipolar major depression (depressive episodes only) or bipolar I disorder (history of manias and depressions) or bipolar II disorder (hypomanias and depressions), current episode depressed acceptable).
3. Must meet criteria for "treatment resistant" depression defined by failure to respond to, or intolerance of, at least 2 treatment trials (antidepressants or ECT) during the current episode.
4. All subjects will be fully ambulatory and in good medical health.
5. Are required to either be antidepressant free for 2 weeks prior to study entry (4 weeks for fluoxetine secondary to long half-life) or be on a fixed psychotropic medication regimen for at least 4 weeks. Subjects and their primary care providers must agree to continue their status (i.e. without antidepressant or on a fixed regimen) until the 12-week assessment is complete.
6. Pre-menopausal female subjects must not be pregnant and must be willing to use adequate contraception during the study period.

Exclusion Criteria:

1. Current or history of psychotic symptoms.
2. Active suicidal ideation (defined as a score of ≥3 on Hamilton Depression Rating Scale (HDRS) suicide item).
3. Prior use of a TNF-alpha antagonist (i.e. etanercept, infliximab, adalimumab) and use of any other immunosuppressant agent (i.e. systemic corticosteroids or anti-proliferative agents such as methotrexate) within one year of study entry.
4. Current use of aspirin, non-steroidal anti-inflammatory agents (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors during the study. Acetaminophen will be allowed.
5. History of any of the following conditions: Congestive heart failure, abnormal electrocardiogram, malignancy, schizophrenia, neurological disease, auto-immune condition (e.g. rheumatoid arthritis, inflammatory bowel disease, multiple sclerosis, lupus), chronic infection (e.g. human immunodeficiency virus, hepatitis B or C), and hematologic, renal or hepatic abnormality.
6. Subjects will be excluded for a positive anti-double stranded DNA antibody test.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H. Miller, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Raison CL, Rutherford RE, Woolwine BJ, Shuo C, Schettler P, Drake DF, Haroon E, Miller AH. A randomized controlled trial of the tumor necrosis factor antagonist infliximab for treatment-resistant depression: the role of baseline inflammatory biomarkers. JAMA Psychiatry. 2013 Jan;70(1):31-41. doi: 10.1001/2013.jamapsychiatry.4. PMID 22945416
- [Result] Weinberger JF, Raison CL, Rye DB, Montague AR, Woolwine BJ, Felger JC, Haroon E, Miller AH. Inhibition of tumor necrosis factor improves sleep continuity in patients with treatment resistant depression and high inflammation. Brain Behav Immun. 2015 Jul;47:193-200. doi: 10.1016/j.bbi.2014.12.016. Epub 2014 Dec 18. PMID 25529904
- [Result] Mehta D, Raison CL, Woolwine BJ, Haroon E, Binder EB, Miller AH, Felger JC. Transcriptional signatures related to glucose and lipid metabolism predict treatment response to the tumor necrosis factor antagonist infliximab in patients with treatment-resistant depression. Brain Behav Immun. 2013 Jul;31:205-15. doi: 10.1016/j.bbi.2013.04.004. Epub 2013 Apr 25. PMID 23624296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Emory University in Atlanta, Georgia. Enrollment began in December 2008 and all participation ended in June 2011.
Pre-assignment Details: Group assignment was stratified based on sex and screening values of C-reactive protein (CRP) concentration (less than 2mg/L or 2mg/L and greater).
Groups:
- Infliximab: Participants receiving 5mg/kg of Infliximab at Baseline, Week 2, and Week 6.
- Placebo: Participants receiving a placebo of normal saline at Baseline, Week 2, and Week 6.
Period: Overall Study
Arm/Group | Infliximab | Placebo
Started | 30 | 30
Completed | 27 | 28
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Schedule conflict | 2 | 0
Not completed — Medical/psychiatric complications | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (8.2) | 44.3 (9.4) | 43.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 23 | 46
  Black | 6 | 5 | 11
  Other | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Hamilton Depression Rating Scale-17 item (HDRS-17) [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Depression Rating Scale-17 item; Minimum score= 0 Maximum score= 54; Higher scores represent greater symptom severity
  scores on a scale | 24.1 (4.0) | 23.6 (3.8) | 23.8 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale 17 (HDRS-17) Scores
Description: The HDRS is a 17-item survey asking respondents to rate the degree of depressive symptoms they are feeling on a scale of 0 to 2-4, where 0 means the symptom is absent and 2-4 means the symptom is very strong. Total scores can range from 0 to 52 where higher scores represent greater symptom severity. Scores of 0-7 are considered normal, scores of 8-16 indicates mild depression, scores of 17-23 indicate moderate depression, and scores of 24 and greater indicate severe depression.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 10 and 12
Population: All participants beginning the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
scores on a scale
  Baseline | 24.1 (4.0) | 23.6 (3.8)
  Week 1 | 20.8 (6.7) | 20.4 (4.9)
  Week 2 | 18.8 (7.0) | 18.3 (6.2)
  Week 4 | 18.8 (6.7) | 16.3 (5.7)
  Week 6 | 17.9 (6.2) | 16.4 (5.9)
  Week 8 | 17.5 (7.4) | 14.8 (6.8)
  Week 10 | 17.4 (8.4) | 13.6 (8.3)
  Week 12 | 16.6 (8.4) | 14.0 (8.1)

2. Secondary Outcome: Number of Participants With a 50% Reduction in Hamilton Depression Rating Scale (HDRS) Scores
Description: The number of participants with a 50% reduction in Hamilton Depression Rating Scale (HDRS) scores at any study point are presented here. The HDRS is a 17-item survey asking respondents to rate the degree of depressive symptoms they are feeling on a scale of 0 to 2-4, where 0 means the symptom is absent and 2-4 means the symptom is very strong. Total scores can range from 0 to 52 where higher scores represent greater symptom severity. Scores of 0-7 are considered normal, scores of 8-16 indicates mild depression, scores of 17-23 indicate moderate depression, and scores of 24 and greater indicate severe depression.
Time Frame: Week 12
Population: All participants beginning the study are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
participants | 15 | 15

3. Secondary Outcome: Number of Remitted Patients During Treatment
Description: The number of participants achieving depression remission are presented here. Depression remission is defined as an HDRS score of ≤7 or a Clinical Global Impression-Improvement (CGI-I) score of 1. The HDRS is a 17-item survey asking respondents to rate the degree of depressive symptoms they are feeling on a scale of 0 to 2-4, where 0 means the symptom is absent and 2-4 means the symptom is very strong. Total scores can range from 0 to 52 where higher scores represent greater symptom severity. Scores of 0-7 are considered normal, scores of 8-16 indicates mild depression, scores of 17-23 indicate moderate depression, and scores of 24 and greater indicate severe depression. The CGI-I scale includes a single item where a health care provider rates the participant's level of clinical improvement on a scale of 1 to 7 where 1 = very much improved since initiation of treatment and 7 = very much worse since initiation of treatment.
Time Frame: Week 12
Population: All participants beginning the study are included in this analysis.
Measure: Number; unit: participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
participants | 9 | 8

4. Secondary Outcome: Inventory of Depressive Symptomatology-Self-Report (IDS-SR) Scores
Description: The Inventory of Depressive Symptomatology-Self-Report (IDS-SR) is a 30-item questionnaire asking respondents about symptoms of depression that they have experienced in the past 7 days. Each item is scored on a 4-point scale where 0 means that the symptom is absent and 3 means that the symptom is very strongly felt. Total scores can range between 0 and 84 and higher scores indicate more severe symptoms of depression.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 10 and 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 43.5 (9.1) | 43.9 (9)
  Week 1 | 37.0 (13) | 38 (12)
  Week 2 | 35.0 (13) | 36 (11)
  Week 4 | 32 (13) | 32 (13)
  Week 6 | 33 (13) | 33 (13)
  Week 8 | 31 (13) | 29 (15)
  Week 10 | 31 (14) | 30 (15)
  Week 12 | 32 (15) | 29 (16)

5. Secondary Outcome: Plasma Concentrations of Interleukin-6 (IL-6)
Description: This study collected blood samples to assess inflammatory markers. IL-6 is a proinflammatory cytokine that is elevated during times of inflammation, infection, illness, and in patients with mood disorders. IL-6 is not present or is low in healthy individuals and exact reference ranges vary by lab, with an example normal reference range of 0.31 to 5.00 picograms per milliliter (pg/mL).
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
pg/ml
  Baseline IL-6 | 2.04 (1.6) | 2.13 (1.19)
  Week 12 IL-6 | 1.88 (2.25) | 1.89 (1.17)

6. Secondary Outcome: Plasma Concentrations of CRP
Description: This study collected blood samples to assess inflammatory markers. CRP increases when inflammation is present and can be measured with a high sensitivity-CRP (hs-CRP) test. Hs-CRP values <1 milligram per liter (mg/L) indicate low inflammation while values >10mg/L indicate inflammation.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 30 | 30
mg/L
  Baseline hs-CRP | 6.21 (9.13) | 5.69 (8.17)
  Week 12 hs-CRP | 3.91 (4.67) | 6.31 (6.92)

7. Secondary Outcome: Plasma Concentrations of Tumor Necrosis Factor (TNF)-Alpha
Description: This study collected blood samples to assess inflammatory markers. Tumor necrosis factor (TNF)-alpha values are invalid due to the administration of infliximab which interferes with the assay procedure.
Time Frame: Baseline, Week 12
Population: TNF-alpha values were invalid due to the administration of infliximab interfering with processing TNF-alpha.
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency is the percentage of time in bed spent sleeping (total sleep time/sleep period time x 100). A sleep efficiency of 80% or greater is considered normal. This outcome measures examines sleep efficiency between study treatment groups.
Time Frame: Baseline, Week 8
Population: This analysis includes participants having complete polysomnography data at baseline and study week 8, and who did not exhibit sleep apnea or periodic limb movement disorder (PLMD).
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 19 | 17
percentage of time asleep
  Baseline | 89.2 (6.7) | 87.9 (10.7)
  Week 8 | 91.5 (7.7) | 90.2 (7.9)

9. Secondary Outcome: Sleep Efficiency in High (CRP>5mg/L) Versus Low (CRP < or =5mg/L) Infliximab-treated Patients
Description: Sleep efficiency is the percentage of time in bed spent sleeping (total sleep time/sleep period time x 100). A sleep efficiency of 80% or greater is considered normal. This outcome measure examines sleep efficiency between participants with high or low baseline CRP.
Time Frame: Baseline, Week 8
Population: This analysis includes participants having complete polysomnography data at baseline and study week 8, who did not exhibit sleep apnea or {LMD, and who were treated with infliximab.
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Groups:
- CRP Greater Than 5 mg/L: Participants with a baseline CRP measurement of greater than 5 mg/L, who were treated with infliximab.
- CRP Less Than or Equal to 5 mg/L: Participants with a baseline CRP measurement of less than or equal to 5 mg/L, who were treated with infliximab.
Arm/Group | CRP Greater Than 5 mg/L | CRP Less Than or Equal to 5 mg/L
Number analyzed (Participants) | 9 | 10
percentage of time asleep
  Baseline | 89.8 (4.2) | 88.6 (8.5)
  Week 8 | 94.5 (3.5) | 88.7 (9.5)

10. Secondary Outcome: Change in Hamilton Depression Rating Scale 17 (HDRS-17) Scores Subgrouped by Baseline Hs-CRP
Description: The effects of baseline high-sensitivity C-reactive protein (hs-CRP) on reduction in depressive symptoms were investigated by examining the least squares mean change in the HDRS score from baseline to week 12 (infliximab minus placebo) among participants with baseline CRP of >1 mg/L, >3 mg/L, and >5 mg/L. A negative change score favors infliximab. The HDRS is a 17-item survey asking respondents to rate the degree of depressive symptoms they are feeling on a scale of 0 to 2-4, where 0 means the symptom is absent and 2-4 means the symptom is very strong. Total scores can range from 0 to 52 where higher scores represent greater symptom severity. Scores of 0-7 are considered normal, scores of 8-16 indicates mild depression, scores of 17-23 indicate moderate depression, and scores of 24 and greater indicate severe depression.
Time Frame: Baseline, Week 12
Population: This analysis includes all study participants in the first group then progressively limits participants in subsequent groups based on baseline hs-CRP concentrations.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- All Participants: All study participants are included.
- Baseline Hs-CRP of >1 mg/L: Participants with a baseline hs-CRP value greater than 1 mg/L.
- Baseline Hs-CRP of > 3: Participants with a baseline hs-CRP value greater than 3 mg/L.
- Baseline Hs-CRP of >5 mg/L: Participants with a baseline hs-CRP value greater than 5 mg/L.
Arm/Group | All Participants | Baseline Hs-CRP of >1 mg/L | Baseline Hs-CRP of > 3 | Baseline Hs-CRP of >5 mg/L
Number analyzed (Participants) | 60 | 45 | 27 | 22
score on a scale | 2.1 (1.8) | 0.3 (2.1) | -1.8 (2.8) | -3.1 (3.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: regular investigator assessment
Groups:
- Placebo: Participants receiving normal saline at Baseline, Week 2, and Week 6.
Arm/Group | Infliximab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=30) | Placebo (N=30)
Headache (Nervous system disorders) | 20 | 18
Coughing (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 6
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Panic attack (Psychiatric disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Increased urinary leukocyte esterase (Renal and urinary disorders) | 0 | 10
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Yeast infection (Infections and infestations) | 3 | 1
Increased urinary white blood cells (Renal and urinary disorders) | 0 | 3
Fever (General disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
This study was underpowered to adequately test placebo response typically reported for treatment resistant depression. Also, no direct measures of the effect of either infliximab or placebo on the central nervous system (CNS) were obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No